CLINICAL TRIAL: NCT04036409
Title: A Randomized Controlled Trial to Assess the Effect of Intensive Blood Pressure Control on Major Cardiovascular Events in Stroke Patients
Brief Title: Optimal Blood Pressure for the prevenTIon of Major vAscuLar Events in Stroke Patients
Acronym: OPTIMAL Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OPTIMAL STROKE Trial
Record Dates: First submitted 2019-07-26; First posted 2019-07-29 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Ischemic Stroke; Blood Pressure; Cognitive Impairment; Vascular Diseases
MeSH Terms: conditions — Ischemic Stroke; Cognitive Dysfunction; Vascular Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive Control of Systolic Blood Pressure (SBP) (Experimental): Participants randomized into the Intensive Blood Pressure arm will have a goal of SBP <120 mm Hg.
  Interventions: Drug: Intensive Control of Systolic Blood Pressure (SBP)
- Standard Control of Systolic Blood Pressure (Active Comparator): Participants randomized into the Standard arm will have a goal of SBP <140 mm Hg
  Interventions: Drug: Standard control of Systolic Blood Pressure (SBP)

INTERVENTIONS:
Drug: Intensive Control of Systolic Blood Pressure (SBP) — Participants in the Intensive arm have a goal of SBP <120 mm Hg. The use of angiotensin converting enzyme (ACE)-inhibitors/Angiotension receptor blockers (ARBs), Thiazide-type diuretics, calcium channel blockers (CCB), Sustained-release calcium channel blockers (CCBs) will be encouraged, preferably fixed-dose combinations of indapamide + perindopril arginine, perindopril arginine + amlodipine or indapamide + perindopril arginine +amlodipine
  Other Names: Intensive BP control targeting SBP <120 mmHg.
  Arms: Intensive Control of Systolic Blood Pressure (SBP)
Drug: Standard control of Systolic Blood Pressure (SBP) — The same medications used in the Intensive BP arm will be used for the Standard BP arm.
  Other Names: Standard control of SBP targeting SBP < 140 mmHg
  Arms: Standard Control of Systolic Blood Pressure

SUMMARY:
Elevated blood pressure (BP) consists of a major public health concern especially in low and middle income countries. Besides being a highly prevalent condition, it is also a risk factor for several major cardiovascular events including stroke (which consists of the second leading cause of death in developing countries) and coronary artery disease, and is also related to cognitive decline. The OPTIMAL Stroke trial consists of a two-arm, multicenter, randomized clinical trial designed to test whether a lower target systolic blood pressure (SBP) as compared to the currently recommended target for stroke patients will reduce the occurrence of major cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* History of ischemic stroke or transient ischemic attack (TIA), considered clinically stable in the 48 hours prior to inclusion in the study. (they will be classified into a recent stroke <120 days or chronic when> 120 days), AND
* Systolic Blood Pressure (SBP) between 130 and 180 mmHg:

  * 130 -180 and use of up to one antihypertensive drug;
  * 130-170 and use of up to two drugs;
  * 130-160 and use of up to three drugs;
  * 130-150 and use of up to four drugs. AND

Exclusion Criteria:

* Severe disability after the event that qualified the patient for the study, defined as a modified Rankin (mRankin) scale equal to or greater than 4.
* Being part of another clinical trial involving interventions for cardiovascular prevention.
* Body mass index > 45 kg/m2.
* Pregnancy or Breastfeeding.
* Secondary hypertension.
* Class IV Canadian Cardiovascular Society (CCS) Resting Angina.
* Acute coronary syndrome in the last six months
* Severe renal dysfunction with GFR < 20 mL/min/1.73m2 calculated by the CKD-EPI equation
* Refusal to consent.
* Symptomatic heart failure - Class IV New York Heart Association (NYHA) or ejection fraction <35% on Doppler echocardiography.
* Conditions that, at the investigators' discretion, limit the patient's participation in the study, including but not limited to the following:

  * Recent history of alcohol and illicit drug abuse.
  * Psychiatric comorbidities (severe depression, schizophrenia, psychosis, etc.).
  * History of poor drug adherence and no attendance at consultations.
  * Planning to change of address in the next four years.
  * Planning to be absent from home city for more than three months in the next year.
  * Residing in the same residence of another patient previously included in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4369 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Time to cardiovascular death, non-fatal myocardial infarction (MI), non-fatal stroke, hospitalization for unstable angina or hospitalization for heart failure [ Time Frame: From randomization; for approximately a median of 3.5 years ] | From randomization; for approximately a median of 3.5 years
  Time to first event of cardiovascular death, non-fatal myocardial infarction (MI), non-fatal stroke, hospitalization for unstable angina or hospitalization for heart failure

SECONDARY OUTCOMES:
Time to cardiovascular death, non-fatal myocardial infarction (MI) or non-fatal stroke [ Time Frame: From randomization; for approximately a median of 3.5 years ] | From randomization; for approximately a median of 3.5 years
  Time to first event of cardiovascular death, non-fatal myocardial infarction (MI) or non-fatal stroke
Time to total death, non-fatal myocardial infarction (MI), non-fatal stroke, hospitalization for unstable angina or hospitalization for heart failure [ Time Frame: From randomization; for approximately a median of 3.5 years ] | From randomization; for approximately a median of 3.5 years
  Time to first event of total death, non-fatal myocardial infarction (MI), non-fatal stroke, hospitalization for unstable angina or hospitalization for heart failure
Time to non-fatal MI, non-fatal stroke, or total death | From randomization; for approximately a median of 3.5 years
  Time to non-fatal MI, non-fatal stroke or total death.
Time to Death | From randomization; for approximately a median of 3.5 years
  Time to all cause death
Time to Renal Death | From randomization; for approximately a median of 3.5 years
  Time to death from renal causes
Time to Renal Outcome | From randomization; for approximately a median of 3.5 years
  Time to Renal Outcome, defined as a 50% reduction in the glomerular filtration rate (GRF) associated with a final GFR of < 60 mL/min/1.73m2 in patients without chronic kidney disease (GFR 60-90 mL/min/1.73m2) at baseline. In those patients with chronic kidney disease (<60 mL/min/1.73m2) at baseline, the renal outcome will be defined as a 50% reduction in GFR or progression of renal disease to stage IV, requiring dialysis or kidney transplantation.
Time to Cardiovascular Death | From randomization; for approximately a median of 3.5 years
  Time to death from cardiovascular causes
Time to Stroke | From randomization; for approximately a median of 3.5 years
  Time to stroke
Time to Hemorrhagic Stroke | From randomization; for approximately a median of 3.5 years
  Time to hemorrhagic stroke
Time to Ischemic Stroke | From randomization; for approximately a median of 3.5 years
  Time to ischemic stroke
Time to Unclassified Stroke | From randomization; for approximately a median of 3.5 years
  Time to unclassified stroke
Time to Transient Ischemic Attack (TIA) | From randomization; for approximately a median of 3.5 years
  Time to Transient Ischemic Attack (TIA)
Time to Myocardial Infarction (MI) | From randomization; for approximately a median of 3.5 years
  Time to myocardial infarction (MI)
Time to Hospitalization due to Heart Failure | From randomization; for approximately a median of 3.5 years
  Time to hospitalization due to heart failure
Time to Hospitalization due to Unstable Angina | From randomization; for approximately a median of 3.5 years
  Time to Hospitalization due to unstable angina
Time to a Composite Outcome of Mild Cognitive Impairment or Probable All Cause Dementia | From randomization; for approximately a median of 3.5 years
  Occurrence of mild cognitive impairment or probable all-cause dementia
Time to Mild Cognitive Impairment | From randomization; for approximately a median of 3.5 years
  Time to Mild Cognitive Impairment
Time to All-Cause Probable Dementia | From randomization; for approximately a median of 3.5 years
  Time to all-cause probable dementia

CONTACTS AND LOCATIONS:
Overall Officials: Otavio Berwanger, MD, PhD, Study Director — Hospital Israelita Albert Einstein
Locations (29):
- Brazil (29):
  - Clínica Silvestre Santé, Rio Branco, Acre
  - Centro de Pesquisas Clinicas (Centro Universitário Cesmac / Hospital do Coração de Alagoas), Maceió, Alagoas
  - Hospital Geral de Fortaleza, Fortaleza, Ceará
  - Universidade Federal do Ceará / Hospital Universitário Walter Cantídio, Fortaleza, Ceará
  - Hospital Universitário Professor Edgard Santos, Salvador, Estado de Bahia
  - Hospital Ana Nery, Salvador, Estado de Bahia
  - Instituto Hospitalar de Base Do Distrito Federal, Brasília, Federal District
  - Universidade Federal de Goias, Goiânia, Goiás
  - Hospital Universitário Maria Aparecida Pedrossian - UFMS, Campo Grande, Mato Grosso do Sul
  - Flumignano Instituto de Medicina, Curitiba, Paraná
  - PROCAPE-Pronto Socorro Cardiológico de PE Prof. Luiz Tavares, Recife, Pernambuco
  - Hospital Moinho de Ventos, Porto Alegre, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital Governador Celso Ramos, Florianópolis, Santa Catarina
  - Clínica Neurológica e Neurocirurgica de Joinville LTDA, Joinville, Santa Catarina
  - CMEP Centro Multidisciplinar de Ensino Especializado e Pesquisa Ltda, Joinville, Santa Catarina
  - Hospital Univ. São Francisco de Assis na Providencia de Deus, Bragança Paulista, São Paulo
  - Universidade Estadual de Campinas - Hospital de Clínicas, Campinas, São Paulo
  - Hospital Carlos Fernando Malzoni, Matão, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto - Universidade de São Paulo, Ribeirão Preto, São Paulo
  - Clínica Vilela e Martin, São José do Rio Preto, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto, São Paulo
  - Irmandade da Santa Casa de Misericórdia de São Paulo, São Paulo, São Paulo
  - UPECLIN - Unidade de Pesquisa Clínica da Faculdade de Medicina de Botucatu - FMB/UNESP, Botucatu
  - Hospital Universitário Pedro Ernesto - UERJ, Rio de Janeiro
  - Hospital das Clínicas da FMUSP, São Paulo
  - Instituto Dante Pazzanese de Cardiologia, São Paulo
  - Hospital São Paulo, São Paulo
  - InCor - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo - HCFMUSP, São Paulo

REFERENCES:
- [Derived] Saiz LC, Gorricho J, Garjon J, Celaya MC, Erviti J, Leache L. Blood pressure targets for the treatment of people with hypertension and cardiovascular disease. Cochrane Database Syst Rev. 2022 Nov 18;11(11):CD010315. doi: 10.1002/14651858.CD010315.pub5. PMID 36398903
- [Derived] Saiz LC, Gorricho J, Garjon J, Celaya MC, Erviti J, Leache L. Blood pressure targets for the treatment of people with hypertension and cardiovascular disease. Cochrane Database Syst Rev. 2020 Sep 9;9(9):CD010315. doi: 10.1002/14651858.CD010315.pub4. PMID 32905623